CLINICAL TRIAL: NCT02016339
Title: Intensive Versus Standard Follow up to Improve Continuous Positive Airway Pressure Compliance: The Greek Experience
Brief Title: Intensive Versus Standard Follow up to Improve Continuous Positive Airway Pressure (CPAP) Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Izolde Bouloukaki, Consultant family physician, Sleep Medicine subspecialty, University of Crete
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPAPCOMPL-01
Record Dates: First submitted 2013-11-27; First posted 2013-12-20 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Standard of Care; Critical Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Active Comparator): 24 hour consultation telephone line to the sleep nurses will be open for the patients. Patients were reviewed at 1 month and at 3 month intervals during the first year and every 6 months thereafter in the CPAP clinic. Additional visits or phone calls by sleep specialist if doubts about a patient's compliance or willingness to continue with the therapy
  Interventions: Behavioral: Standard care
- Intensive care (Active Comparator): Standard group care plus:
  Involvement of the patient's partner or family. Extra education on sleep apnea syndrome and CPAP by sleep specialists via a 15-min videotape. 10- to 15-min lecture from the sleep clinic's nurses. Phone calls by nurses at 2 and 7 days. Early review of patients by sleep specialists at 15 and 30 days. Home visits by sleep nurses, if there doubts about a patients adherence.
  Interventions: Behavioral: Intensive care

INTERVENTIONS:
Behavioral: Standard care — 24-h consultation telephone line to the sleep nurses to answer questions regarding CPAP usage. Patients were reviewed at 1 month and at 3 month intervals during the first year and every 6 months thereafter in the CPAP clinic by the nurse. Additional visits or phone calls by sleep specialist if doubts about a patient's compliance or willingness to continue with the therapy.
  Arms: Standard Care
Behavioral: Intensive care — Standard group care plus: Involvement of the patient's partner or family necessary. Extra education on sleep apnea and CPAP by sleep specialists via a 15-min videotape. 10- to 15-min lecture from the sleep clinic's nurses after CPAP titration study. Phone calls by nurses at 2 and 7 days. Early review of patients by sleep specialists at 15 and 30 days. Home visits by sleep nurses, if there doubts about a patients adherence
  Arms: Intensive care

SUMMARY:
The purpose of this study was to compare the effects on sleepiness, quality of life, depression, hospitalization and deaths rate, of intensive vs standard interventions, on CPAP adherence, 2 years after CPAP initiation.

DETAILED DESCRIPTION:
There is limited data concerning long-term randomized clinical trials proving the long-term efficacy of intensive use, follow programs on improving CPAP use. Therefore the investigators aimed to compare the effects on sleepiness, quality of life, depression, hospitalization and deaths rate, of intensive vs standard interventions, on CPAP adherence, 2 years after CPAP initiation.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed obstructive sleep apnea syndrome by polysomnography according to standard criteria,
* with moderate to severe sleep apnea,
* no history of previously CPAP therapy and
* with an above-elementary school education.

Exclusion Criteria:

* refusal to participate,
* refusal to CPAP therapy,
* previous CPAP treatment,
* central sleep apnoea syndrome,
* Cheyne-stokes breathing pattern,
* obesity hypoventilation syndrome,
* restrictive ventilator syndromes,
* congestive heart failure,
* history of life-threatening arrhythmias,
* cardiomyopathy,
* long term oxygen therapy,
* family or personal history of mental illness,
* with drug or alcohol abuse,
* severe cognitive impairment,
* concurrent oncologic diseases and
* history of narcolepsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2836 (Actual)
Dates: Start 2007-06; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Effect of intensive intervention on CPAP adherence | 24 months

SECONDARY OUTCOMES:
Effect of intensive intervention on sleepiness. | 24 months
Effect of intensive intervention on mood. | 24 months
Effect of intensive intervention on quality of life | 24 months

OTHER OUTCOMES:
Effect of intensive intervention on hospitalization rate. | 24 months
Effect of intensive intervention on withdrawal of CPAP | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sophia E Schiza, MD, PhD, Study Chair — University of Crete; Charalampos Mermigkis, MD, PhD, Study Director — Sleep Disorders Center, Pulmonary Department, 401 General Army Hospital, Athens, Greece; Izolde Bouloukaki, MD, PhD, Principal Investigator — University of Crete

REFERENCES:
- [Derived] Bouloukaki I, Giannadaki K, Mermigkis C, Tzanakis N, Mauroudi E, Moniaki V, Michelakis S, Siafakas NM, Schiza SE. Intensive versus standard follow-up to improve continuous positive airway pressure compliance. Eur Respir J. 2014 Nov;44(5):1262-74. doi: 10.1183/09031936.00021314. Epub 2014 Jul 3. PMID 24993911